CLINICAL TRIAL: NCT06129175
Title: Cytopeutics® A Phase II-III Double-Blind Randomized Controlled Study to Assess the Efficacy of Umbilical Cord Mesenchymal Stem Cells (Neuroncell-EX) Transplantation in Patients With Acute Ischemic Stroke
Brief Title: UCMSCs as Treatment for Patients With Acute Ischemic Stroke (Stroke Neuroncell-EX)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cytopeutics Sdn. Bhd. (Industry)
Collaborators: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: POD0031/CP/R
Record Dates: First submitted 2023-10-12; First posted 2023-11-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Mesenchymal stem cells
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuroncell-EX (Experimental): Umbilical cord-derived mesenchymal stem cells
  Interventions: Biological: Neuroncell-EX
- Control (Placebo Comparator): Normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Neuroncell-EX — Intravenous infusion of Neuroncell-EX (2 million UCMSCs per kg body weight) on day 1 and day 14 plus standard medical care.
  Arms: Neuroncell-EX
Other: Placebo — Intravenous infusion of Placebo (normal saline) on day 1 and day 14 plus standard medical care.
  Arms: Control

SUMMARY:
The primary objective of this study is to evaluate the functional recovery based on Barthel index (BI) and modified Rankin Scale (mRS) while the secondary objectives are to assess the survival and re-admission rate as well as to investigate the inflammatory response in a subclinical study within 1 year of Neuroncell-EX infusion in participants with acute ischemic stroke.

DETAILED DESCRIPTION:
Background: Ischemic stroke is a serious cerebrovascular disease with high morbidity and disability worldwide. Despite the great efforts that have been made, the prognosis of stroke patients remains unsatisfactory. Mesenchymal stem cells (MSCs) therapy is an emerging treatment studied in various medical conditions including autoimmune, inflammatory as well as central nervous system diseases. The mechanism of MSCs in the treatment of ischemic stroke involved with immune regulation, neuroprotection, angiogenesis, and neural circuit reconstruction. A large number of preclinical data have proved the feasibility of MSCs in the treatment of stroke where the administration of MSCs can alleviate neurological deficits. Similarly, a number of clinical trials have also proved the effectiveness and safety of MSCs in the treatment of stroke. Among these is a phase 2, single-center, assessor-blinded randomized controlled study by investigators using bone marrow-derived MSCs in patients with subacute middle cerebral artery infarct. The investigators demonstrated the safety, tolerability, and efficacy of intravenous infusion of MSCs with significant improvement in median infarct volume (Law et al., 2021).

Objective: To determine the efficacy of intravenous infusion of allogeneic Cytopeutics umbilical cord mesenchymal stem cells (Neuroncell-EX) in participants with acute ischemic stroke.

Study Design: This is a phase II-III double-blind randomized controlled study involving 80 participants, diagnosed with acute ischemic stroke admitted to HCTM-UKM. Investigational treatment arm (Group A-MSCs) consist of 40 participants will receive Neuroncell-EX whereas control treatment arm (Group B-Control) consist of 40 participants will receive placebo. Both groups will also receive standard medical care for acute stroke. Efficacy assessments will include Barthel index (BI) and modified Rankin Scale (mRS), Functional Magnetic Resonance Imaging (fMRI) and blood tests including biomarkers within 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be aged ≥ 18 years old.
2. Patients with acute ischemic stroke symptom onset within 4 weeks.
3. Patients diagnosed with "moderate to severe" based on NIHSS (6-24) at the time of recruitment.
4. Patients who are not eligible for thrombolysis or thrombectomy.
5. Written informed consent by the patient or next-of-kin.

Exclusion Criteria:

1. Patients who are medically unfit such as those who are haemodynamically unstable or whose general condition is deteriorating.
2. Patients with transient ischemic attack (TIA).
3. Patients who have been diagnosed with malignancy (past or present) or primary haematological disorders.
4. Patients who have renal impairment with serum creatinine more than 200 µmol/l or creatinine clearance less than 30 ml/min.
5. Patients who have liver impairment with serum aspartate transaminase (AST) and alanine aminotransferase (ALT) two times greater than upper normal limit.
6. Patients who are pregnant or are breastfeeding.
7. Patients diagnosed with brain hemorrhage or other pathological brain disorders such as vascular malformation (brain arteriovenous malformation), tumor, abscess, cardiogenic, inflammatory and infectious cerebral embolism or other common non- ischemic brain diseases, or diagnosed with severe brain atrophy, as determined by CT or MRI scans.
8. Patients diagnosed/suspected diagnosis with acute coronary syndrome.
9. Patients with congestive cardiac failure.
10. Patients with history of confirmed or suspected pulmonary embolism or chronic obstructive pulmonary disease (COPD).
11. Patients with mental, cognitive or psychological disorders that affects their understanding and adherence to research procedures and follow-ups.
12. Patients that are undergoing experimental drug or instrument testing or have participated in other clinical drug trials in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Barthel Index (BI) | Baseline, 6 weeks, 3 months, 6 months and 12 months
  Functional recovery after stroke onset is measured by the Barthel Index (BI). BI score from 0-100, higher scores mean better outcome. The investigators measure and compare the BI score for ischemic stroke patients who received Neuroncell-EX and control treatments.
Modified Rankin Scale | Baseline, 6 weeks, 3 months, 6 months and 12 months
  Functional recovery after stroke onset is measured by the modified Rankin Scale (mRS). mRS is a 7 point (0-6) ranking scale to assess neurological disability. A score of 0 indicates normal functions with no symptoms while higher scores indicates more severe neurological disability.The investigators measure and compare the mRS score for ischemic stroke patients who received Neuroncell-EX and control treatments.

SECONDARY OUTCOMES:
Number of participants with adverse events due to umbilical cord-derived mesenchymal stem cells infusion as assessed by clinical examination. | Baseline, day 1, day 14, 6 weeks, 3 months, 6 months and 12 months
  Presence or absence of any adverse events due to the umbilical cord-derived mesenchymal stem cells (UC-MSCs) infusion, sepsis, organ failure (clinically apparent or subclinical), hospitalization, cancers and death during the study period based on clinical examination.
Survival and Re-admission rate | Baseline, day 1, day 14, 6 weeks, 3 months, 6 months and 12 months
  Survival and re-admission rate
Blood inflammatory markers before and after umbilical cord derived mesenchymal stem cell infusion based on subclinical analysis. | Baseline, 6 months and 12 months
  Biomarkers concentration: Interleukin-6 (IL-6), interleukin-2 (IL-2), matrix metalloproteinase-9 (MMP-9), tumour necrosis factor alpha (TNFα), interleukin-1beta (IL-1β), vascular endothelial growth factor (VEGF), interleukin-10 (IL-10), Interleukin-1 receptor antagonist protein (IL-1Ra) and transforming growth factor beta 1 (TGF-β1).

CONTACTS AND LOCATIONS:
Overall Officials: Wan Nur Nafisah Wan Yahya, Principal Investigator — National University of Malaysia
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No